CLINICAL TRIAL: NCT04954079
Title: Retrograde Approach in Ambulatory Practice
Acronym: RAAR
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Other Study IDs: RAAR
Record Dates: First submitted 2021-06-29; First posted 2021-07-08 (Actual); Last update posted 2023-08-09 (Actual); Status verified 2023-08

CONDITIONS: Obliterative Arterial Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Obliterative arterial disease of the lower limbs affects 200 million people worldwide, including approximately 40 million in Europe. This disease is associated with a significant increase in morbidity and mortality.

The most common clinical symptomatology is difficulty walking (intermittent claudication). Less frequent but more severe, critical ischemia includes rest pain requiring analgesics, and trophic disorders (ulcers, gangrene), which may lead to amputation. The Rutherford classification groups the different clinical forms of this pathology. The classic risk factors of cardiovascular pathologies, such as age, smoking, hypertension, diabetes and hypercholesterolemia, are closely linked to Obliterative arterial disease of the lower limbs. Over the past 20 years, the interventional management of this condition has undergone a paradigm shift. The rise of endovascular surgery has broadened the range of therapeutic possibilities, while reducing the impact on patients. Advances in equipment and imaging quality have made it possible to treat increasingly complex lesions, allowing this type of technique to be offered to patients initially treated with conventional surgery (Trans-Atlantic Inter-Society Consensus (TASC) C and D). Unfortunately, for long recanalizations and calcified lesions, the crossing of the lesion and its re-entry into the true arterial lumen is a failure in 25% of cases. It is with this in mind that retrograde puncture and the associated SAFARI (Subintimal Arterial Flossing with Anterograde-retrograde Intervention) technique were developed. In case of failure to cross the lesion by anterograde, intraluminal or subintimal, a retrograde puncture downstream, echo or radio guided, is performed. The vessels most often punctured are the popliteal artery or the leg axes. Recanalization of the lesion is done by retrograde approach. The guidewire introduced distally is recovered in the introducer through which the first recanalization attempt was made. The procedure is then performed in the classical way using the anterograde approach. At the end of the procedure, hemostasis of the puncture site is obtained by prolonged inflation of a balloon or the placement of a covered stent. Initially reserved for critically ischemic patients (Rutherford 4-6), this technique tends to be extended to claudicant patients (Rutherford 2-3). Zhuang et al have recently demonstrated the efficacy and safety of this technique in a large cohort of patients.

In parallel with the evolution of revascularization techniques, the evolution of care pathways has given ambulatory care a prominent place. Since January 2020, in the vascular surgery department of GHPSJ, peripheral angioplasties are mostly performed on an outpatient basis. The patients treated are classified as Rutherford 2 to 5 in most cases. No adverse events related to this management have been reported. To date, no study evaluating the feasibility and safety of retrograde punctures in the outpatient setting has been performed.

ELIGIBILITY:
Inclusion Criteria:

* Patient with age ≥ 18 years
* Patient with symptomatic AOMI (Rutherford 2 to 6) with indication for revascularization
* Patient with ambulatory management
* Patient whose management requires retrograde arterial puncture
* Francophone patient
* Patient who does not object to the use of his/her data for this research

Exclusion Criteria:

* Patient under guardianship or curatorship
* Patient deprived of liberty
* Patient under court protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: These patients are referred for endovascular revascularization of lower extremity obliterative arterial disease, Rutherford stage 2 to 6, between 01/06/2021 and 01/06/2022.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2021-07-21 (Actual); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-08-31 (Estimated)

PRIMARY OUTCOMES:
Serious adverse event | Month 1
  This outcome corresponds to the number of the serious adverse event on the operated limb.

CONTACTS AND LOCATIONS:
Overall Officials: Maxime Raux, MD, Principal Investigator — Fondation Hôpital Saint-Joseph
Locations (2):
- France (2):
  - Centre Hospitalier Universitaire de Brest, Brest
  - Groupe Hospitalier Paris Saint-Joseph, Paris

REFERENCES:
- [Background] Aboyans V, Ricco JB, Bartelink MEL, Bjorck M, Brodmann M, Cohnert T, Collet JP, Czerny M, De Carlo M, Debus S, Espinola-Klein C, Kahan T, Kownator S, Mazzolai L, Naylor AR, Roffi M, Rother J, Sprynger M, Tendera M, Tepe G, Venermo M, Vlachopoulos C, Desormais I; ESC Scientific Document Group. 2017 ESC Guidelines on the Diagnosis and Treatment of Peripheral Arterial Diseases, in collaboration with the European Society for Vascular Surgery (ESVS): Document covering atherosclerotic disease of extracranial carotid and vertebral, mesenteric, renal, upper and lower extremity arteriesEndorsed by: the European Stroke Organization (ESO)The Task Force for the Diagnosis and Treatment of Peripheral Arterial Diseases of the European Society of Cardiology (ESC) and of the European Society for Vascular Surgery (ESVS). Eur Heart J. 2018 Mar 1;39(9):763-816. doi: 10.1093/eurheartj/ehx095. No abstract available. PMID 28886620
- [Background] Fowkes FG, Rudan D, Rudan I, Aboyans V, Denenberg JO, McDermott MM, Norman PE, Sampson UK, Williams LJ, Mensah GA, Criqui MH. Comparison of global estimates of prevalence and risk factors for peripheral artery disease in 2000 and 2010: a systematic review and analysis. Lancet. 2013 Oct 19;382(9901):1329-40. doi: 10.1016/S0140-6736(13)61249-0. Epub 2013 Aug 1. PMID 23915883
- [Background] Sampson UK, Fowkes FG, McDermott MM, Criqui MH, Aboyans V, Norman PE, Forouzanfar MH, Naghavi M, Song Y, Harrell FE Jr, Denenberg JO, Mensah GA, Ezzati M, Murray C. Global and regional burden of death and disability from peripheral artery disease: 21 world regions, 1990 to 2010. Glob Heart. 2014 Mar;9(1):145-158.e21. doi: 10.1016/j.gheart.2013.12.008. PMID 25432124